CLINICAL TRIAL: NCT02288247
Title: A Randomized, Double Blind, Placebo-Controlled, Phase IIIb Study of the Efficacy and Safety of Continuing Enzalutamide in Chemotherapy Naïve Metastatic Castration Resistant Prostate Cancer Patients Treated With Docetaxel Plus Prednisolone Who Have Progressed on Enzalutamide Alone
Brief Title: A Study to Assess the Benefit of Treatment Beyond Progression With Enzalutamide in Men Who Are Starting Treatment With Docetaxel After Worsening of Their Prostate Cancer When Taking Enzalutamide Alone
Acronym: PRESIDE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Europe Ltd. (Industry)
Collaborators: Medivation LLC, a wholly owned subsidiary of Pfizer Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 9785-MA-1001; 2013-004711-50 (EudraCT Number)
Record Dates: First submitted 2014-11-07; First posted 2014-11-11 (Estimated); Results first posted 2021-12-15 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
Keywords: Metastatic; Castration-resistant; Docetaxel; Chemotherapy- Naïve; Enzalutamide; Prostate Cancer; Chemotherapy Naïve Metastatic Castration Resistant Prostate Cancer; Prednisolone; Xtandi; Metastatic Castration Resistant Prostate Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms | interventions — enzalutamide; Docetaxel; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Enzalutamide (Experimental): Participants (Pts) received OL enzalutamide 160 mg QD from Day 1 in Period 1 (P1) until they were either randomized to Period 2 (P2), were ineligible, experienced intolerable toxicity, withdrew, or died. Pts with confirmed disease progression in P1, meeting eligibility, were randomized to receive placebo/enzalutamide 160 mg QD with docetaxel 75 mg/m^2 in 1hour infusion every 3 weeks & prednisolone 5mg twice daily in P2. Docetaxel & prednisolone were administered for upto 10 cycles (1 cycle=3 weeks) or more per investigator discretion, while placebo/enzalutamide continued until progression, toxicity, withdrawal, or death. Extension(EXT) phase was available for Pts in P1& P2 who were not meeting primary endpoint. Enzalutamide continued until disease progression, intolerable toxicity, withdrawal, or death. Pts not entering EXT discontinued and received local care. Those benefiting from enzalutamide in EXT at study closure continued in study 9785-CL-0123 or via commercial enzalutamide.
  Interventions: Drug: Enzalutamide; Drug: Docetaxel; Drug: Prednisolone
- Placebo (Placebo Comparator): Participants received an OL treatment with enzalutamide 160 mg capsules, orally once daily from day 1 in period 1 until randomization to period 2 treatment, confirmation of ineligibility for period 2 treatment, intolerable toxicity, withdrawal, or death, whichever occurred first. Participants with confirmed disease progression on enzalutamide in period 1 and who continued to meet all eligibility criteria received placebo matched to enzalutamide, orally once daily in combination with docetaxel 75 mg/m^2 in a one-hour infusion every 3 weeks and prednisolone 5 mg orally twice daily, DB in period 2. Docetaxel and prednisolone were administered up to 10 cycles (1 cycle = 3 weeks) or additional cycles as assessed by the investigator and enzalutamide was administered until disease progression, intolerable toxicity, withdrawal or death, whichever occurred first. Participants discontinued the study and received local standard of care.
  Interventions: Drug: Docetaxel; Drug: Prednisolone; Drug: Placebo

INTERVENTIONS:
Drug: Enzalutamide — Oral
  Other Names: Xtandi; ASP9785
  Arms: Enzalutamide
Drug: Docetaxel — intravenous infusion
Drug: Prednisolone — Oral
Drug: Placebo — Oral
  Arms: Placebo

SUMMARY:
The purpose of the study was to understand if there was benefit in continued treatment with a medicine called enzalutamide, when starting treatment with docetaxel and prednisolone (a standard chemotherapy for prostate cancer), after the prostate cancer had gotten worse when treated with enzalutamide alone.

DETAILED DESCRIPTION:
The study was conducted in consecutive periods of open label treatment with enzalutamide followed by randomized double-blind treatment with continued enzalutamide or placebo, in combination with docetaxel and prednisolone.

Open Label (Period 1)

Participants received open label treatment (OL) with enzalutamide. At week 13, all participants were assessed by prostate-specific antigen (PSA) and imaging. Participants with no confirmed PSA response or evidence of radiographic progression were ineligible for participation in Period 2 and typically had safety follow up; however, Period 1 treatment continued for some participants as long as the investigator considered it to be of clinical benefit (stopping on initiation of any new antineoplastic therapy). Participants with confirmed PSA response continued Period 1 until disease progression.

Enrollment to Period 2 ceased after approximately 274 participants had been enrolled or 182 primary endpoint events had been reached, whichever occurred first. Participants who were not randomized into period 2 at this time continued to receive open label treatment in an extension period.

Randomization (Double Blind [DB]) (Period 2)

Participants with confirmed disease progression on enzalutamide alone who continued to meet all eligibility criteria proceeded to randomization. Treatment allocation was in a 1:1 ratio, stratified by disease progression in Period 1 to the following treatments:

* Enzalutamide with docetaxel and prednisolone
* Placebo with docetaxel and prednisolone

Any ongoing participants in Period 2 at the point of unblinding in the enzalutamide+docetaxel arm that were still receiving and benefitting from enzalutamide treatment, had the option to continue treatment via an extension period.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features;
* Ongoing androgen deprivation therapy (ADT) with a luteinizing hormone-releasing hormone (LHRH) agonist or antagonist at a stable dose and schedule within 4 weeks of initiation of investigational medicinal product (IMP), or bilateral orchiectomy (i.e., surgical or medical castration);
* Metastatic disease documented by at least 2 bone lesions on bone scan, or soft tissue disease documented by computed tomography (CT)/magnetic resonance imaging (MRI);
* Progressive disease at study entry defined as the following occurring in the setting of castrate levels of testosterone: Prostate specific antigen (PSA) progression defined by a minimum of three rising PSA levels with an interval of ≥ 1 week between each determination.
* Asymptomatic or minimally symptomatic prostate cancer (Brief Pain Inventory - Short Form (BPI-SF) question 3 score of < 4);
* Eastern Cooperative Oncology Group (ECOG) performance score of 0-1;
* Estimated life expectancy of ≥ 12 months;
* Be suitable and willing to receive chemotherapy as part of the trial;
* Able to swallow the IMP and comply with study requirements;
* Subject agreed not to participate in another interventional study while on treatment.

Exclusion Criteria:

* Prior treatment with the following agents for the treatment of prostate cancer: Aminoglutethimide; Ketoconazole; Abiraterone; Enzalutamide or participation in a clinical trial of enzalutamide; 223Ra, 89Sr, 153Sm, 186Re/188Re; Immunomodulatory therapies; Cytotoxic chemotherapy; Participation in a clinical trial of an investigational agent that inhibits the AR or androgen synthesis unless the treatment was placebo;
* Current or prior treatment within 4 weeks prior to initiation of investigational medicinal product (IMP) with the following agents for the treatment of prostate cancer: Antiandrogens; 5-α reductase inhibitors; Estrogens; Anabolic steroids; Drugs with antiandrogenic properties; Progestational agents;
* Subject had received investigational therapy within 28 days or 5 half-lives whichever was longer, prior to initiation of IMP;
* Use of opiate analgesia for pain from prostate cancer within 4 weeks prior to initiation of IMP;
* Radiation therapy to bone lesions or prostatic bed within 4 weeks prior to initiation of IMP;
* Major surgery within 4 weeks prior to initiation of IMP;
* History of seizure or any condition that may predispose to seizures at any time in the past. History of loss of consciousness or transient ischemic attack within 12 months prior to Screening;
* Known or suspected brain metastasis or active leptomeningeal disease;
* History of another malignancy within the previous 5 years other than non-melanoma skin cancer;
* Clinically significant cardiovascular disease;
* Gastrointestinal disorders affecting absorption;
* Medical contraindications to the use of prednisolone or docetaxel;
* Allergies to any of the active ingredients or excipients in the study drugs

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 688 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2024-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Europe Ltd.
Locations (89):
- Austria (2):
  - Site AT43004, Linz
  - Site AT43001, Vienna
- Belgium (3):
  - Site BE32003, Bonheiden
  - Site BE32002, Liège
  - Site BE32004, Ottignies
- Czechia (4):
  - Site CZ42004, Brno
  - Site CZ42003, Olomouc
  - Site CZ42002, Plzeň -Lochotín
  - Site CZ42001, Prague
- France (9):
  - Site FR33012, Albi
  - Site FR33003, Montpellier
  - Site FR33002, Nîmes
  - Site FR33008, Paris
  - Site FR33014, Paris
  - Site FR33004, Plérin
  - Site FR33013, Quimper
  - Site FR33011, Reims
  - Site FR33005, Suresnes
- Germany (10):
  - Site DE49018, Nürtingen, Baden-Wurttemberg
  - Site DE49008, Aachen
  - Site DE49010, Bergisch Gladbach
  - Site DE49001, Hanover
  - Site DE49006, Heidelberg
  - Site DE49003, Mannheim
  - Site DE49002, Münster
  - Site DE49015, Tübingen
  - Site DE49017, Ulm
  - Site DE49004, Wuppertal
- Greece (5):
  - Site GR30001, Heraklion, Crete
  - Site GR30004, Heraklion, Crete
  - Site GR30003, Athens
  - Site GR30006, Athens
  - Site GR30005, Thessaloniki
- Italy (8):
  - Site IT39001, Arezzo
  - Site IT39012, Brescia
  - Site IT39003, Milan
  - Site IT39008, Naples
  - Site IT39010, Pavia
  - Site IT39005, Roma
  - Site IT39004, Rome
  - Site IT39002, Terni
- Netherlands (5):
  - Site NL31002, Amsterdam
  - Site NL31007, Blaricum
  - Site NL31004, Hoofddorp
  - Site NL31010, Nieuwegein
  - Site NL31003, Rotterdam
- Norway (3):
  - Site NO47005, Drammen
  - Site NO47001, Kristiansand
  - Site NO47004, Stavanger
- Poland (5):
  - Site PL48004, Gdansk
  - Site PL48003, Krakow
  - Site PL48002, Lodz
  - Site PL48006, Warsaw
  - Site PL48005, Warsaw
- Russia (6):
  - Site RU70004, Obninsk, Kaluga Oblast
  - Site RU70002, Moscow
  - Site RU70001, Moscow
  - Site RU70003, Moscow
  - Site RU70005, Saint Petersburg
  - Site RU70006, Saint Petersburg
- Spain (10):
  - Site ES34005, Lugo
  - Site ES34003, Madrid
  - Site ES34001, Madrid
  - Site ES34002, Madrid
  - Site ES34010, Madrid
  - Site ES34007, Málaga
  - Site ES34009, Murcia
  - Site ES34008, Santander
  - Site ES34004, Seville
  - Site ES34006, Valencia
- Sweden (4):
  - Site SE46002, Gothenburg
  - Site SE46005, Kalmar
  - Site SE46003, Solna
  - Site SE46004, Uppsala
- Switzerland (2):
  - Site CH41005, Locarno, Canton Ticino
  - Site CH41009, Zurich
- Turkey (Türkiye) (3):
  - Site TR90001, Ankara
  - Site TR90003, Istanbul
  - Site TR90002, Izmir
- United Kingdom (10):
  - Site GB44010, Aberdeen
  - Site GB44004, Cambridge
  - Site GB44018, Cardiff
  - Site GB44014, Exeter
  - Site GB44003, London
  - Site GB44007, Metropolitan Borough of Wirral
  - Site GB44020, Northwood
  - Site GB44015, Norwich
  - Site GB44002, Nottingham
  - Site GB44017, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Merseburger AS, Attard G, Astrom L, Matveev VB, Bracarda S, Esen A, Feyerabend S, Senkus E, Lopez-Brea Piqueras M, Boysen G, Gourgioti G, Martins K, Chowdhury S. Continuous enzalutamide after progression of metastatic castration-resistant prostate cancer treated with docetaxel (PRESIDE): an international, randomised, phase 3b study. Lancet Oncol. 2022 Nov;23(11):1398-1408. doi: 10.1016/S1470-2045(22)00560-5. Epub 2022 Oct 18. PMID 36265504
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14680&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male participants with metastatic Castration-Resistant Prostate Cancer (mCRPC) who had progressed while on luteinizing hormone-releasing hormone (LHRH) agonist/antagonist or after receiving a bilateral orchiectomy and had not yet received chemotherapy were enrolled in the study.
Pre-assignment Details: Following Screening, participants received open-label (OL) treatment with enzalutamide in period 1 followed by period 2 randomized double-blind (DB) treatment with continued enzalutamide or placebo, adding with docetaxel and prednisolone. Participants were stratified by disease progression in Period 1 (evidence of radiographic progression or not).
Groups:
- Enzalutamide: Participants received OL enzalutamide 160 milligrams (mg) capsules orally once daily (QD) from Day 1 in Period (P) 1 until they were either randomized to P2 treatment, deemed ineligible, experienced intolerable toxicity, withdrew, or died, whichever came first. Participants with confirmed disease progression on enzalutamide in Period 1 who continued to meet eligibility criteria, were randomized to receive either placebo or enzalutamide 160 mg capsules orally QD with docetaxel 75 milligrams per meter square (mg/m^2) in 1-hour infusion every 3 weeks and prednisolone 5 mg orally twice daily in DB P2. Docetaxel and prednisolone were administered for up to 10 cycles (1 cycle = 3 weeks) or additional cycles as determined by investigator, while placebo/enzalutamide was continued until disease progression, intolerable toxicity, withdrawal, or death whichever occurred first. An Extension (EXT) phase was available for participants still in P1 and participants in P2 not meeting the primary endpoint, when the data cut-off for analysis was reached. Treatment with enzalutamide continued until the disease progression, intolerable toxicity, participant withdrawal or death. Participants who did not enter EXT phase had discontinued study and received local standard of care treatment. Those who were still benefiting from enzalutamide treatment in EXT phase at study closure continued enzalutamide therapy in another Astellas-sponsored study 9785-CL-0123 or via commercially available enzalutamide.
- Placebo: Participants received an OL treatment with enzalutamide 160 mg capsules, orally once daily from day 1 in P1 until randomization to P2 treatment, confirmation of ineligibility for P2 treatment, intolerable toxicity, withdrawal, or death, whichever occurred first. Participants with confirmed disease progression on enzalutamide in P1 and who continued to meet all eligibility criteria received placebo matched to enzalutamide, orally once daily in combination with docetaxel 75 mg/m^2 in a one-hour infusion every 3 weeks and prednisolone 5 mg orally twice daily, DB in P2. Docetaxel and prednisolone were administered up to 10 cycles (1 cycle = 3 weeks) or additional cycles as assessed by the investigator and enzalutamide was administered until disease progression, intolerable toxicity, withdrawal or death, whichever occurred first. Participants discontinued the study and received local standard of care.
Period: Period 1: OL Treatment (Max: 462 Weeks)
Arm/Group | Enzalutamide | Placebo
Started | 688 | 0
Treated | 687 | 0
Completed (Completed participants are those who did not have a treatment discontinuation.) | 0 | 0
Not Completed | 688 | 0
Not completed — Adverse Event | 52 | 0
Not completed — Death | 35 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Progressive Disease | 393 | 0
Not completed — Protocol Violation | 9 | 0
Not completed — Withdrawal by Subject | 54 | 0
Not completed — Other | 142 | 0
Not completed — Study Terminated By Sponsor | 2 | 0
Period: Period 2: DB Treatment (Max: 180 Weeks)
Arm/Group | Enzalutamide | Placebo
Started | 137 (137 participants from period 1 were randomized to period 2.) | 136 (136 participants from period 1 were randomized to period 2.)
Treated | 136 | 135
Completed | 0 | 1
Not Completed | 137 | 135
Not completed — Adverse Event | 10 | 8
Not completed — Death | 8 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Progressive Disease | 87 | 94
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 7 | 7
Not completed — Other | 21 | 21
Not completed — Randomized but not treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set 1 (SAF1) included all participants who received at least one dose of investigational medicinal product (IMP) in period 1.
Groups:
- Enzalutamide: Participants received OL enzalutamide 160 mg capsules orally QD from Day 1 in Period 1 until they were either randomized to Period 2 treatment, deemed ineligible, experienced intolerable toxicity, withdrew, or died, whichever came first. Participants with confirmed disease progression on enzalutamide in Period 1, who continued to meet eligibility criteria, were randomized to receive either placebo or enzalutamide 160 mg capsules orally QD with docetaxel 75 mg/m^2 in 1-hour infusion every 3 weeks and prednisolone 5 mg orally twice daily in DB Period 2. Docetaxel and prednisolone were administered for up to 10 cycles (1 cycle = 3 weeks) or additional cycles as determined by investigator, while placebo/enzalutamide was continued until disease progression, intolerable toxicity, withdrawal, or death whichever occurred first. An EXT was available for patients still in P1 and patients in P2 not meeting the primary endpoint, when the data cut-off for analysis was reached. Treatment with enzalutamide continued until the disease progression, intolerable toxicity, participant withdrawal or death. Participants who did not enter extension phase had discontinued study and received local standard of care treatment. Those who were still benefiting from enzalutamide treatment in EXT phase at study closure continued enzalutamide therapy in another Astellas-sponsored study 9785-CL-0123 or via commercially available enzalutamide.
Arm/Group | Enzalutamide
Number analyzed (Participants) | 687
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 687
Race/Ethnicity, Customized [Number; unit: participants]
  Race : White | 681
  Race : Black Or African American | 5
  Race : Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS: time from randomization (Period 2 Week 1) to earliest progression event. Progression is defined as radiographic progression, unequivocal clinical progression, or death on study. Radiographic progression is defined for bone disease by appearance of ≥ 2 new lesions on whole-body radionuclide bone scan per Prostate Cancer Clinical Trials Working Group 2 (PCWG2) criteria (i.e., unconfirmed progressive disease) that needs to be confirmed in the next assessment (i.e., progressive disease in the next assessment) or for soft tissue disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Unequivocal clinical progression is defined as new onset cancer pain requiring chronic administration of opiate analgesia or deterioration from prostate cancer of Eastern Cooperative Oncology Group (ECOG) performance status score to ≥ 3, or initiation of subsequent lines of cytotoxic chemotherapy or radiation therapy or surgical intervention due to complications of tumor progression.
Time Frame: From date of randomization to the earliest of either documented disease progression (median duration: 35 weeks)
Population: The Full Analysis Set (FAS) consisted of all participants who were randomized and received at least one dose of IMP.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Enzalutamide: Participants with confirmed disease progression on enzalutamide in period 1 and who continued to meet all eligibility criteria received enzalutamide 160 mg capsules, orally once daily in combination with docetaxel 75 mg/m^2 in a one-hour infusion every 3 weeks and prednisolone 5 mg orally twice daily, in DB treatment period 2. Docetaxel and prednisolone were administered up to 10 cycles (1 cycle= 3 weeks) or additional cycles as assessed by the investigator and enzalutamide was administered until disease progression, intolerable toxicity, withdrawal or death, whichever occurred first. Participants could continue the extension period if they were still receiving study drug in Period 1 when enrollment to Period 2 closed or when the data cut-off for analysis was reached in Period 2, until the investigator or participant decided to stop or disease progression, intolerable toxicity, withdrawal or death, whichever occurred first.
- Placebo: Participants with confirmed disease progression on enzalutamide in period 1 and who continued to meet all eligibility criteria received placebo matched to enzalutamide, orally once daily in combination with docetaxel 75 mg/m^2 in a one-hour infusion every 3 weeks and prednisolone 5 mg orally twice daily, in DB treatment period 2. Docetaxel and prednisolone were administered up to 10 cycles (1 cycle= 3 weeks) or additional cycles as assessed by the investigator and enzalutamide was administered until disease progression, intolerable toxicity, withdrawal or death, whichever occurred first. Participants could continue the extension period if they were still receiving study drug in Period 1 when enrollment to Period 2 closed or when the data cut-off for analysis was reached in Period 2, until the investigator or participant decided to stop or disease progression, intolerable toxicity, withdrawal or death, whichever occurred first.
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 136 | 135
months | 9.53 [8.25 to 10.87] | 8.28 [6.28 to 8.71]
Statistical Analysis 1: Comparison: Enzalutamide vs Placebo; Test type: Superiority; p = 0.027, Cox proportional hazards model — From the Cox proportional hazards model with covariates for treatment and disease progression in Period 1 (radiographic, nonradiographic); Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.53 to 0.96]

2. Secondary Outcome: Time to Prostate-specific Antigen (PSA) Progression
Description: Time to PSA progression, defined as the time from randomization (Period 2 Week 1) to the date of the first PSA value in Period 2 demonstrating progression (Period 2). The PSA progression date is defined as the date that a ≥ 25% increase and an absolute increase of ≥ 2 ng/mL above the nadir recorded in Period 2 is documented, which must be confirmed by a second consecutive value obtained at least 3 weeks later.
Time Frame: From date of randomization to the first PSA value (median duration: 35 weeks)
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 136 | 135
months | 8.44 [8.18 to 9.00] | 6.24 [5.42 to 8.31]
Statistical Analysis 1: Comparison: Enzalutamide vs Placebo; Test type: Superiority; p = 0.002, Cox proportional hazards model — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.41 to 0.82]

3. Secondary Outcome: Prostate-specific Antigen (PSA) Response
Description: PSA response, defined as a decrease in percentage change from randomization (Period 2 Week 1) of 50% or more. PSA response was derived at Week 13 and at any time after randomization in Period 2. PSA response at any time is defined as a decrease in percentage change from randomization (Period 2 Week 1) at any time after randomization of 50% or more. Percentage of participants with PSA response was reported.
Time Frame: Randomization, Week 13, any time after randomization in Period 2 (median of 35 weeks)
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 136 | 135
percentage of participants
  Week 13 | 44.9 | 25.2
  Any time after randomization (median of 35 weeks) | 55.9 | 37.0

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR, defined as the best overall radiographic response after randomization (Period 2 Week 1) as per Investigator assessments of response for soft tissue disease per RECIST 1.1, in participants who had a measurable tumor. ORR was reported as the percentage of participants with complete response (CR) or partial response (PR). CR was defined as disappearance of all target and nontarget lesions. Any pathological lymph nodes (whether target or nontarget) must have reduction in short axis to < 10 mm from baseline measurement. PR was defined as at least a 30% decrease in the sum of diameters (longest for nonnodal lesions, short axis for nodal lesions) of target lesions taking as reference to the baseline sum of diameters.
Time Frame: From date of randomization up to median duration of 35 weeks
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 136 | 135
percentage of participants | 31.6 [0.60 to 0.76] | 25.9 [0.66 to 0.81]
Statistical Analysis 1: Comparison: Enzalutamide vs Placebo; Test type: Superiority; p = 0.142, Cochran-Mantel-Haenszel — From the Cochran-Mantel-Haenszel test stratified by disease progression (radiographic, non-radiographic) in Period 1

5. Secondary Outcome: Time to Pain Progression
Description: The time to an increase of >=30% from randomization (Period 2 Week 1) in average BPI-SF item scores (items 3, 4, 5, 6) at two consecutive evaluations >=3 weeks apart without decrease in analgesic score according to the World health Organization (WHO). Only participants with an average pain intensity item score >=4 were considered. The BPI-SF was an instrument to document pain-related functional impairment and contains 7 questions which included pain intensity [(items 3, 4, 5 and 6): worst pain, least pain, average pain and current pain, with scales from 0 (no pain) to 10 (pain as bad as you can imagine)] and pain interference ](items 9A to 9G): general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life, with scales from 0 (does not interfere) to 10 (completely interferes)]. The BPI-SF total score for pain intensity was calculated as the mean of the 4 scores for the 4 items of pain intensity.
Time Frame: From date of randomization up to median duration of 35 weeks
Population: Data was not estimable as none of the participants met the criteria for pain progression
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Time to Opiate Use for Cancer-related Pain
Description: Time to opiate use for cancer-related pain, defined as the time from randomization (Period 2 Week 1) to initiation of chronic administration of opiate analgesia [parenteral opiate use for ≥7 days or use of WHO Analgesic Ladder Level 3 oral opiates for ≥3 weeks].
Time Frame: From date of randomization up to median duration of 35 weeks
Population: Data was not estimable as none of the participants had cancer-related pain.
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Time to First Skeletal-related Event (SRE)
Description: Time to first SRE, defined as the time from randomization (Period 2 Week 1) to radiation therapy or surgery to bone, pathologic bone fracture, spinal cord compression, or change of antineoplastic therapy to treat bone pain.
Time Frame: From date of randomization up to median duration of 35 weeks
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 136 | 135
months | 21.98 [15.18 to NA] — Upper limit of 95% confidence interval was not estimable due to insufficient number of events. | 17.35 [17.35 to NA] — Upper limit of 95% confidence interval was not estimable due to insufficient number of events.
Statistical Analysis 1: Comparison: Enzalutamide vs Placebo; Test type: Superiority; p = 0.994, Cox proportional hazards model — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.47 to 2.13]

8. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy - Prostate (FACT-P)
Description: FACT-P quality of life questionnaire is a multi-dimensional, self-reported quality of life instrument specifically designed for use with prostate cancer participants. It consists of 27 core items which assess participant function in four domains rated on 0 to 4 Likert-type scale: physical well-being (PWB) (7 items; 0 [worst] to 4 [better], score range 0-28), social/family well-being (SWB) (7 items; 0 [worst] to 4 [better], score range 0-28), emotional well-being (EWB) (6 items; 0 [worst] to 4 [better], score range 0-24), and functional well-being (FWB) (7 items; 0 [worst] to 4 [better], score range 0-28), which is further supplemented by 12 site-specific items to assess for prostate-related symptoms (Prostate Cancer Subscale [PCS] 12 items rated on Likert-type scale 0 [worst] to 4 [better], score range 0-48). The total domain scores and PCS subscale score are then combined to a global quality of life score ranging between 0 to 156; higher scores representing better quality of life.
Time Frame: Period 2: Baseline, weeks 1, 13, 25, 37, 49, 61, 73, 85, 97, 109, 121, 133, 145, 157, 169, 181
Population: Participants in the FAS population with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 124 | 133
score on a scale
  EWB: Baseline: number analyzed (Participants) | 122 | 132
  EWB: Baseline | 0.00 (0.00) | 0.00 (0.00)
  EWB: Change at Week 1: number analyzed (Participants) | 104 | 115
  EWB: Change at Week 1 | 0.00 (0.00) | 0.00 (0.00)
  EWB: Change at Week 13: number analyzed (Participants) | 88 | 99
  EWB: Change at Week 13 | 1.15 (4.15) | 1.36 (3.63)
  EWB: Change at Week 25: number analyzed (Participants) | 60 | 64
  EWB: Change at Week 25 | 0.69 (3.85) | 1.03 (3.58)
  EWB: Change at Week 37: number analyzed (Participants) | 55 | 45
  EWB: Change at Week 37 | 1.91 (3.85) | 1.43 (3.73)
  EWB: Change at Week 49: number analyzed (Participants) | 38 | 22
  EWB: Change at Week 49 | 1.22 (3.62) | 0.73 (4.24)
  EWB: Change at Week 61: number analyzed (Participants) | 18 | 6
  EWB: Change at Week 61 | 0.59 (4.52) | 2.00 (3.58)
  EWB: Change at Week 73: number analyzed (Participants) | 11 | 1
  EWB: Change at Week 73 | 1.69 (3.13) | -1.00
  EWB: Change at Week 85: number analyzed (Participants) | 5 | 1
  EWB: Change at Week 85 | 1.00 (4.06) | -5.00
  EWB: Change at Week 97: number analyzed (Participants) | 4 | 0
  EWB: Change at Week 97 | 3.90 (4.75) |
  EWB: Change at Week 109: number analyzed (Participants) | 3 | 0
  EWB: Change at Week 109 | 2.93 (3.49) |
  EWB: Change at Week 121: number analyzed (Participants) | 2 | 0
  EWB: Change at Week 121 | 4.00 (2.83) |
  EWB: Change at Week 133: number analyzed (Participants) | 2 | 0
  EWB: Change at Week 133 | 2.00 (0.00) |
  EWB: Change at Week 145: number analyzed (Participants) | 1 | 0
  EWB: Change at Week 145 | 2.00 |
  EWB: Change at Week 157: number analyzed (Participants) | 1 | 0
  EWB: Change at Week 157 | 2.00 |
  EWB: Change at Week 169: number analyzed (Participants) | 1 | 0
  EWB: Change at Week 169 | 1.00 |
  EWB: Change at Week 181: number analyzed (Participants) | 1 | 0
  EWB: Change at Week 181 | 2.00 |
  FWB: Baseline: number analyzed (Participants) | 122 | 132
  FWB: Baseline | 0.0000 (0.0000) | 0.0000 (0.0000)
  FWB: Change at Week 1: number analyzed (Participants) | 104 | 115
  FWB: Change at Week 1 | 0.0000 (0.0000) | 0.0000 (0.0000)
  FWB: Change at Week 13: number analyzed (Participants) | 88 | 99
  FWB: Change at Week 13 | -1.8144 (5.0586) | -0.3121 (4.7437)
  FWB: Change at Week 25: number analyzed (Participants) | 60 | 64
  FWB: Change at Week 25 | -2.4472 (5.2508) | -0.8229 (5.2563)
  FWB: Change at Week 37: number analyzed (Participants) | 55 | 45
  FWB: Change at Week 37 | -1.5697 (6.3251) | -0.1459 (3.2857)
  FWB: Change at Week 49: number analyzed (Participants) | 38 | 22
  FWB: Change at Week 49 | -1.1579 (6.7284) | -1.3818 (4.5238)
  FWB: Change at Week 61: number analyzed (Participants) | 18 | 6
  FWB: Change at Week 61 | 0.0000 (4.7651) | -2.3333 (2.8048)
  FWB: Change at Week 73: number analyzed (Participants) | 11 | 1
  FWB: Change at Week 73 | -1.8182 (3.5726) | -2.0000
  FWB: Change at Week 85: number analyzed (Participants) | 5 | 1
  FWB: Change at Week 85 | 1.2000 (4.8166) | 0.0000
  FWB: Change at Week 97: number analyzed (Participants) | 4 | 0
  FWB: Change at Week 97 | -0.5000 (1.7321) |
  FWB: Change at Week 109: number analyzed (Participants) | 3 | 0
  FWB: Change at Week 109 | -1.3333 (3.2146) |
  FWB: Change at Week 121: number analyzed (Participants) | 2 | 0
  FWB: Change at Week 121 | -1.5000 (0.7071) |
  FWB: Change at Week 133: number analyzed (Participants) | 2 | 0
  FWB: Change at Week 133 | -0.5000 (2.1213) |
  FWB: Change at Week 145: number analyzed (Participants) | 1 | 0
  FWB: Change at Week 145 | -2.0000 |
  FWB: Change at Week 157: number analyzed (Participants) | 1 | 0
  FWB: Change at Week 157 | 0.0000 |
  FWB: Change at Week 169: number analyzed (Participants) | 1 | 0
  FWB: Change at Week 169 | -1.0000 |
  FWB: Change at Week 181: number analyzed (Participants) | 1 | 0
  FWB: Change at Week 181 | 0.0000 |
  Global Score: Baseline: number analyzed (Participants) | 121 | 129
  Global Score: Baseline | 0.0000 (0.0000) | 0.0000 (0.0000)
  Global Score: Change at Week 1: number analyzed (Participants) | 104 | 113
  Global Score: Change at Week 1 | 0.0000 (0.0000) | 0.0000 (0.0000)
  Global Score: Change at Week 13: number analyzed (Participants) | 84 | 95
  Global Score: Change at Week 13 | -0.7836 (17.7356) | 1.7986 (16.3294)
  Global Score: Change at Week 25: number analyzed (Participants) | 58 | 61
  Global Score: Change at Week 25 | -5.9204 (18.2107) | 1.0762 (17.0168)
  Global Score: Change at Week 37: number analyzed (Participants) | 52 | 43
  Global Score: Change at Week 37 | -1.5351 (20.3721) | 0.1649 (15.8335)
  Global Score: Change at Week 49: number analyzed (Participants) | 37 | 21
  Global Score: Change at Week 49 | -4.4880 (24.6865) | -4.6202 (17.9530)
  Global Score: Change at Week 61: number analyzed (Participants) | 17 | 6
  Global Score: Change at Week 61 | -0.2957 (17.6915) | 6.0939 (8.8208)
  Global Score: Change at Week 73: number analyzed (Participants) | 11 | 0
  Global Score: Change at Week 73 | -0.3917 (18.3346) |
  Global Score: Change at Week 85: number analyzed (Participants) | 5 | 0
  Global Score: Change at Week 85 | 1.7636 (11.7476) |
  Global Score: Change at Week 97: number analyzed (Participants) | 4 | 0
  Global Score: Change at Week 97 | 6.2864 (9.8128) |
  Global Score: Change at Week 109: number analyzed (Participants) | 3 | 0
  Global Score: Change at Week 109 | -2.7333 (17.6299) |
  Global Score: Change at Week 121: number analyzed (Participants) | 1 | 0
  Global Score: Change at Week 121 | 4.0000 |
  Global Score: Change at Week 133: number analyzed (Participants) | 2 | 0
  Global Score: Change at Week 133 | -7.0000 (4.2426) |
  Global Score: Change at Week 145: number analyzed (Participants) | 1 | 0
  Global Score: Change at Week 145 | -11.0000 |
  Global Score: Change at Week 157: number analyzed (Participants) | 1 | 0
  Global Score: Change at Week 157 | -1.0000 |
  Global Score: Change at Week 169: number analyzed (Participants) | 1 | 0
  Global Score: Change at Week 169 | -10.0000 |
  Global Score: Change at Week 181: number analyzed (Participants) | 1 | 0
  Global Score: Change at Week 181 | -4.0000 |
  PWB: Baseline | 0.0000 (0.0000) | 0.0000 (0.0000)
  PWB: Change at Week 1: number analyzed (Participants) | 106 | 115
  PWB: Change at Week 1 | 0.0000 (0.0000) | 0.0000 (0.0000)
  PWB: Change at Week 13: number analyzed (Participants) | 90 | 100
  PWB: Change at Week 13 | -1.3322 (6.0823) | -0.6347 (4.4643)
  PWB: Change at Week 25: number analyzed (Participants) | 62 | 65
  PWB: Change at Week 25 | -3.1317 (6.5208) | -0.4590 (4.2887)
  PWB: Change at Week 37: number analyzed (Participants) | 56 | 45
  PWB: Change at Week 37 | -2.1786 (5.5611) | -0.9556 (4.3691)
  PWB: Change at Week 49: number analyzed (Participants) | 38 | 23
  PWB: Change at Week 49 | -2.5316 (8.0882) | -1.3913 (6.1625)
  PWB: Change at Week 61: number analyzed (Participants) | 18 | 6
  PWB: Change at Week 61 | -1.3889 (6.9886) | 1.3333 (3.8297)
  PWB: Change at Week 73: number analyzed (Participants) | 11 | 1
  PWB: Change at Week 73 | -0.3636 (8.0408) | 3.0000
  PWB: Change at Week 85: number analyzed (Participants) | 5 | 1
  PWB: Change at Week 85 | 1.0000 (10.3682) | 3.0000
  PWB: Change at Week 97: number analyzed (Participants) | 4 | 0
  PWB: Change at Week 97 | 1.7500 (10.4363) |
  PWB: Change at Week 109: number analyzed (Participants) | 3 | 0
  PWB: Change at Week 109 | -0.6667 (13.6504) |
  PWB: Change at Week 121: number analyzed (Participants) | 2 | 0
  PWB: Change at Week 121 | -4.0000 (1.4142) |
  PWB: Change at Week 133: number analyzed (Participants) | 2 | 0
  PWB: Change at Week 133 | -4.5000 (0.7071) |
  PWB: Change at Week 145: number analyzed (Participants) | 1 | 0
  PWB: Change at Week 145 | -4.0000 |
  PWB: Change at Week 157: number analyzed (Participants) | 1 | 0
  PWB: Change at Week 157 | 0.0000 |
  PWB: Change at Week 169: number analyzed (Participants) | 1 | 0
  PWB: Change at Week 169 | -4.0000 |
  PWB: Change at Week 181: number analyzed (Participants) | 1 | 0
  PWB: Change at Week 181 | -2.0000 |
  PCS: Baseline: number analyzed (Participants) | 123 | 130
  PCS: Baseline | 0.0000 (0.0000) | 0.0000 (0.0000)
  PCS: Change at Week 1: number analyzed (Participants) | 106 | 113
  PCS: Change at Week 1 | 0.0000 (0.0000) | 0.0000 (0.0000)
  PCS: Change at Week 13: number analyzed (Participants) | 86 | 95
  PCS: Change at Week 13 | 1.1842 (6.1843) | 1.6011 (6.0731)
  PCS: Change at Week 25: number analyzed (Participants) | 60 | 63
  PCS: Change at Week 25 | -0.4775 (6.2665) | 1.8632 (6.3433)
  PCS: Change at Week 37: number analyzed (Participants) | 53 | 44
  PCS: Change at Week 37 | -1.1433 (7.3006) | 0.6988 (7.1353)
  PCS: Change at Week 49: number analyzed (Participants) | 37 | 22
  PCS: Change at Week 49 | -1.8465 (8.6083) | -0.7223 (7.8442)
  PCS: Change at Week 61: number analyzed (Participants) | 17 | 6
  PCS: Change at Week 61 | 0.3690 (6.0031) | 4.2606 (3.1148)
  PCS: Change at Week 73: number analyzed (Participants) | 11 | 0
  PCS: Change at Week 73 | 0.9174 (7.8001) |
  PCS: Change at Week 85: number analyzed (Participants) | 5 | 0
  PCS: Change at Week 85 | 2.1636 (5.6123) |
  PCS: Change at Week 97: number analyzed (Participants) | 4 | 0
  PCS: Change at Week 97 | 3.8864 (3.3380) |
  PCS: Change at Week 109: number analyzed (Participants) | 3 | 0
  PCS: Change at Week 109 | -1.6667 (5.8595) |
  PCS: Change at Week 121: number analyzed (Participants) | 1 | 0
  PCS: Change at Week 121 | 2.0000 |
  PCS: Change at Week 133: number analyzed (Participants) | 2 | 0
  PCS: Change at Week 133 | -3.0000 (4.2426) |
  PCS: Change at Week 145: number analyzed (Participants) | 1 | 0
  PCS: Change at Week 145 | -5.0000 |
  PCS: Change at Week 157: number analyzed (Participants) | 1 | 0
  PCS: Change at Week 157 | 0.0000 |
  PCS: Change at Week 169: number analyzed (Participants) | 1 | 0
  PCS: Change at Week 169 | -3.0000 |
  PCS: Change at Week 181: number analyzed (Participants) | 1 | 0
  PCS: Change at Week 181 | -2.0000 |
  SWB: Baseline | 0.0000 (0.0000) | 0.0000 (0.0000)
  SWB: Change at Week 1: number analyzed (Participants) | 106 | 115
  SWB: Change at Week 1 | 0.0000 (0.0000) | 0.0000 (0.0000)
  SWB: Change at Week 13: number analyzed (Participants) | 90 | 100
  SWB: Change at Week 13 | -0.1581 (4.1893) | -0.2953 (5.0738)
  SWB: Change at Week 25: number analyzed (Participants) | 62 | 65
  SWB: Change at Week 25 | -0.3634 (5.6959) | -0.0462 (3.7933)
  SWB: Change at Week 37: number analyzed (Participants) | 56 | 45
  SWB: Change at Week 37 | 0.8798 (4.6897) | -0.3963 (3.3279)
  SWB: Change at Week 49: number analyzed (Participants) | 38 | 23
  SWB: Change at Week 49 | -0.0719 (6.2561) | -0.7536 (4.3164)
  SWB: Change at Week 61: number analyzed (Participants) | 18 | 6
  SWB: Change at Week 61 | -0.8167 (3.3323) | 0.8333 (5.7067)
  SWB: Change at Week 73: number analyzed (Participants) | 11 | 1
  SWB: Change at Week 73 | -0.8182 (2.7863) | -24.0000
  SWB: Change at Week 85: number analyzed (Participants) | 5 | 1
  SWB: Change at Week 85 | -3.6000 (3.7815) | -24.0000
  SWB: Change at Week 97: number analyzed (Participants) | 4 | 0
  SWB: Change at Week 97 | -2.7500 (5.8523) |
  SWB: Change at Week 109: number analyzed (Participants) | 3 | 0
  SWB: Change at Week 109 | -2.0000 (4.3589) |
  SWB: Change at Week 121: number analyzed (Participants) | 2 | 0
  SWB: Change at Week 121 | 0.5000 (0.7071) |
  SWB: Change at Week 133: number analyzed (Participants) | 2 | 0
  SWB: Change at Week 133 | -1.0000 (1.4142) |
  SWB: Change at Week 145: number analyzed (Participants) | 1 | 0
  SWB: Change at Week 145 | -2.0000 |
  SWB: Change at Week 157: number analyzed (Participants) | 1 | 0
  SWB: Change at Week 157 | -3.0000 |
  SWB: Change at Week 169: number analyzed (Participants) | 1 | 0
  SWB: Change at Week 169 | -3.0000 |
  SWB: Change at Week 181: number analyzed (Participants) | 1 | 0
  SWB: Change at Week 181 | -2.0000 |

9. Secondary Outcome: Change From Baseline in EuroQOL 5-dimension 5-level Questionnaire [EQ-5D-5L] Visual Analog Scale (VAS)
Description: The EQ-5D-5L VAS records the participant's self-rated health on a vertical visual analogue scale, where the endpoints are labelled from 0 (worst health imaginable) to 100 (best health imaginable).
Time Frame: Period 2: Baseline, weeks 1, 13, 25, 37, 49, 61, 73, 85, 97, 109, 121, 133, 145, 157, 169, 181
Population: Participants in the FAS population with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enzalutamide | Placebo
Number analyzed (Participants) | 121 | 130
score on a scale
  Baseline | 0.0 (0.0) | 0.0 (0.0)
  Change at Week 1: number analyzed (Participants) | 106 | 113
  Change at Week 1 | 0.0 (0.0) | 0.0 (0.0)
  Change at Week 13: number analyzed (Participants) | 89 | 100
  Change at Week 13 | 2.3 (19.7) | -0.8 (17.8)
  Change at Week 25: number analyzed (Participants) | 63 | 64
  Change at Week 25 | -3.0 (18.6) | -0.2 (17.7)
  Change at Week 37: number analyzed (Participants) | 55 | 47
  Change at Week 37 | -1.3 (21.7) | 0.4 (15.8)
  Change at Week 49: number analyzed (Participants) | 42 | 24
  Change at Week 49 | -2.5 (25.7) | -8.3 (23.3)
  Change at Week 61: number analyzed (Participants) | 19 | 6
  Change at Week 61 | 1.3 (22.6) | 2.5 (25.2)
  Change at Week 73: number analyzed (Participants) | 11 | 1
  Change at Week 73 | -3.5 (30.8) | -20.0
  Change at Week 85: number analyzed (Participants) | 5 | 1
  Change at Week 85 | 7.2 (20.7) | -10.0
  Change at Week 97: number analyzed (Participants) | 4 | 0
  Change at Week 97 | 17.8 (27.0) |
  Change at Week 109: number analyzed (Participants) | 3 | 0
  Change at Week 109 | 17.7 (23.6) |
  Change at Week 121: number analyzed (Participants) | 2 | 0
  Change at Week 121 | -7.0 (4.2) |
  Change at Week 133: number analyzed (Participants) | 2 | 0
  Change at Week 133 | 0.5 (13.4) |
  Change at Week 145: number analyzed (Participants) | 1 | 0
  Change at Week 145 | 1.0 |
  Change at Week 157: number analyzed (Participants) | 1 | 0
  Change at Week 157 | -4.0 |
  Change at Week 169: number analyzed (Participants) | 1 | 0
  Change at Week 169 | 2.0 |
  Change at Week 181: number analyzed (Participants) | 1 | 0
  Change at Week 181 | -4.0 |

ADVERSE EVENTS:
Time Frame: From first dose up to 71 weeks
Description: Safety Analysis Set 1 (SAF1) consisted of all participants who took at least one dose of study drug during Period 1. Safety Analysis Set 2 (SAF2) consisted of all participants who took at least one dose of study drug during Period 2.
Groups:
- Period 1: Enzalutamide: Participants received OL enzalutamide 160 mg capsules orally QD from Day 1 in Period 1 until they were either randomized to Period 2 treatment, deemed ineligible, experienced intolerable toxicity, withdrew, or died, whichever came first. An EXT phase was available for participants still in P1 not meeting the primary endpoint, when the data cut-off for analysis was reached. Treatment with enzalutamide continued until the disease progression, intolerable toxicity, participant withdrawal or death. Participants who did not enter EXT phase had discontinued study and received local standard of care treatment. Those who were still benefiting from enzalutamide treatment in EXT phase at study closure continued enzalutamide therapy in another Astellas-sponsored study 9785-CL-0123 or via commercially available enzalutamide.
- Period 2: Enzalutamide: Participants with confirmed disease progression on enzalutamide in P1 and who continued to meet all eligibility criteria received enzalutamide 160 mg capsules, orally once daily in combination with docetaxel 75 mg/m^2 in a one-hour infusion every 3 weeks and prednisolone 5 mg orally twice daily, DB treatment in P2. Docetaxel and prednisolone were administered up to 10 cycles (1 cycle= 3 weeks) or additional cycles as assessed by the investigator and enzalutamide was administered until disease progression, intolerable toxicity, withdrawal or death, whichever occurred first. An EXT was available for participants in P2 not meeting the primary endpoint, when the data cut-off for analysis was reached. Treatment with enzalutamide continued until the disease progression, intolerable toxicity, participant withdrawal or death. Participants who did not enter EXT phase had discontinued study and received local standard of care treatment. Those who were still benefiting from enzalutamide treatment in EXT phase at study closure continued enzalutamide therapy in another Astellas-sponsored study 9785-CL-0123 or via commercially available enzalutamide.
- Period 2: Placebo: Participants with confirmed disease progression on enzalutamide in P1 and who continued to meet all eligibility criteria received placebo matched to enzalutamide, orally once daily in combination with docetaxel 75 mg/m^2 in a one-hour infusion every 3 weeks and prednisolone 5 mg orally twice daily, DB in P2. Docetaxel and prednisolone were administered up to 10 cycles (1 cycle= 3 weeks) or additional cycles as assessed by the investigator and enzalutamide was administered until disease progression, intolerable toxicity, withdrawal or death, whichever occurred first.
Arm/Group | Period 1: Enzalutamide | Period 2: Enzalutamide | Period 2: Placebo
All-Cause Mortality (participants affected / at risk) | 51/687 | 18/136 | 15/135
Serious Adverse Events (participants affected / at risk) | 238/687 | 67/136 | 52/135
Other Adverse Events (participants affected / at risk) | 523/687 | 125/136 | 123/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Enzalutamide (N=687) | Period 2: Enzalutamide (N=136) | Period 2: Placebo (N=135)
Anaemia (Blood and lymphatic system disorders) | 9 (17) | 3 (3) | 2 (2)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 10 (10) | 15 (17)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 11 (21) | 5 (12)
Pancytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 4 (4) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 12 (14) | 3 (3) | 2 (2)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 6 (6) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Dressler's syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 9 (10) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Blindness (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Exfoliation glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 5 (7) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (3) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Asthenia (General disorders) | 2 (2) | 2 (2) | 0 (0)
Chest pain (General disorders) | 4 (5) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 4 (4) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 5 (6) | 1 (1) | 3 (4)
Generalised oedema (General disorders) | 0 (0) | 1 (2) | 1 (1)
Hypothermia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 5 (6) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 6 (7) | 2 (2)
Sudden death (General disorders) | 2 (2) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Catheter bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dacryocystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infective aneurysm (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 2 (3) | 0 (0)
Lyme disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Meningitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 5 (6) | 3 (3)
Peritonitis (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 4 (4) | 3 (3)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 5 (5) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Streptococcal urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection pseudomonal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 6 (7) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 8 (9) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 6 (7) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Incorrect dose administered (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Urostomy complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 1 (1) | 0 (0) | 0 (0)
General physical condition abnormal (Investigations) | 5 (8) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (3) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Troponin I increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (3) | 1 (1) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (14) | 2 (2) | 3 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (5) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant neoplasm of pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 22 (24) | 6 (6) | 6 (6)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Soft tissue sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Uveal melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Brain compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 5 (5) | 1 (1) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0)
Hemiplegia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Motor dysfunction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Paraplegia (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 6 (6) | 5 (5) | 1 (1)
Syncope (Nervous system disorders) | 5 (5) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vascular dementia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 3 (3) | 0 (0) | 0 (0)
Thrombosis in device (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 7 (8) | 2 (2) | 2 (2)
Bladder outlet obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder tamponade (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 12 (17) | 1 (1) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 6 (7) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Urethral obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 1 (2) | 0 (0) | 1 (1)
Urinary bladder polyp (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 7 (7) | 0 (0) | 1 (1)
Urinary tract disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Scrotal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 2 (2) | 1 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bone operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cardiac pacemaker removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Carpal tunnel decompression (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Catheterisation venous (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Arterial insufficiency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Malignant hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Enzalutamide (N=687) | Period 2: Enzalutamide (N=136) | Period 2: Placebo (N=135)
Anaemia (Blood and lymphatic system disorders) | 49 (63) | 27 (47) | 15 (32)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 11 (37) | 16 (48)
Neutropenia (Blood and lymphatic system disorders) | 5 (5) | 41 (125) | 43 (129)
Lacrimation increased (Eye disorders) | 2 (3) | 25 (28) | 6 (7)
Constipation (Gastrointestinal disorders) | 60 (64) | 12 (21) | 15 (17)
Diarrhoea (Gastrointestinal disorders) | 63 (77) | 37 (51) | 42 (67)
Nausea (Gastrointestinal disorders) | 69 (79) | 26 (33) | 25 (31)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 5 (5) | 8 (9)
Vomiting (Gastrointestinal disorders) | 22 (25) | 8 (8) | 6 (6)
Asthenia (General disorders) | 109 (175) | 46 (94) | 35 (64)
Fatigue (General disorders) | 159 (194) | 40 (65) | 28 (41)
Mucosal inflammation (General disorders) | 3 (3) | 10 (14) | 17 (19)
Oedema peripheral (General disorders) | 26 (31) | 16 (18) | 20 (23)
Pyrexia (General disorders) | 18 (19) | 9 (11) | 7 (9)
Nasopharyngitis (Infections and infestations) | 28 (33) | 4 (5) | 8 (8)
Fall (Injury, poisoning and procedural complications) | 47 (64) | 6 (7) | 4 (4)
Haemoglobin decreased (Investigations) | 15 (17) | 2 (3) | 7 (7)
Neutrophil count decreased (Investigations) | 3 (4) | 7 (14) | 7 (27)
Weight decreased (Investigations) | 30 (36) | 11 (11) | 2 (2)
White blood cell count decreased (Investigations) | 9 (12) | 5 (17) | 7 (24)
Decreased appetite (Metabolism and nutrition disorders) | 69 (86) | 23 (28) | 17 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 70 (85) | 25 (27) | 10 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 117 (153) | 13 (15) | 14 (15)
Bone pain (Musculoskeletal and connective tissue disorders) | 64 (80) | 12 (14) | 14 (16)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 33 (38) | 5 (7) | 7 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 22 (23) | 9 (9) | 7 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 44 (55) | 7 (10) | 7 (7)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 23 (26) | 8 (12) | 11 (14)
Dizziness (Nervous system disorders) | 45 (49) | 5 (5) | 6 (6)
Dysgeusia (Nervous system disorders) | 10 (12) | 18 (22) | 9 (9)
Headache (Nervous system disorders) | 44 (56) | 5 (6) | 8 (10)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 22 (29) | 12 (21)
Paraesthesia (Nervous system disorders) | 22 (24) | 8 (10) | 10 (21)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 12 (16) | 14 (25)
Taste disorder (Nervous system disorders) | 7 (7) | 6 (6) | 9 (11)
Haematuria (Renal and urinary disorders) | 41 (50) | 4 (5) | 7 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 27 (32) | 11 (15) | 10 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 28 (30) | 11 (13) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 13 (16) | 7 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 44 (56) | 37 (48)
Dry skin (Skin and subcutaneous tissue disorders) | 14 (14) | 12 (12) | 5 (5)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 13 (13) | 7 (8)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (9) | 2 (3)
Nail toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 11 (16) | 5 (7)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 13 (14) | 12 (16)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 10 (15) | 1 (1)
Hot flush (Vascular disorders) | 73 (89) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 91 (103) | 3 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT02288247/Prot_002.pdf
  • Statistical Analysis Plan (2024-01-23): https://cdn.clinicaltrials.gov/large-docs/47/NCT02288247/SAP_003.pdf